CLINICAL TRIAL: NCT06487104
Title: Safety, Feasibility, and Impact on Pulmonary Secretion Management Comparing the Use of TrachPhone and External Humidifier After Tracheostomy
Brief Title: Use of TrachPhone in Tracheostomized Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TrachPhone
Record Dates: First submitted 2024-04-05; First posted 2024-07-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Tracheostomy
Keywords: Heat and Moisture Exchangers; Secretion

STUDY DESIGN:
Intervention Model Description: Single-center, two-armed randomized controlled trial with a subsequent feasibility phase, transitioning control-group patients to investigational device arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - HME (Experimental): 24/7 use of TrachPhone HME for the entirety of study
  Interventions: Device: TrachPhone HME
- Arm 2 - EH (Active Comparator): 24/7 use of EH until first follow-up (T1), then 24/7 use of TrachPhone HME for the remainder of the study participation.
  Interventions: Device: TrachPhone HME; Device: External Humidifier (Usual Care)

INTERVENTIONS:
Device: TrachPhone HME — Use of TrachPhone HME for humidification of inhaled air in tracheostomized patients.
  The TrachPhone HME is an HME specifically designed for tracheostomy patients.
Device: External Humidifier (Usual Care) — Usual care routines using an External Humidifier for humidification of inhaled air in tracheostomized patients.
  Arms: Arm 2 - EH

SUMMARY:
The use of Heat and Moisture Exchangers (HMEs) and their positive impact on pulmonary health have been extensively studied in patients with head and neck cancer but have not been systematically explored in other patient populations breathing through a neck stoma.

The objective of this clinical investigation is to compare the use of HMEs to the use of External Humidifiers (EHs) on pulmonary secretion management, their usability and safety, for humidifying inhaled air in patients that received a tracheostomy due to a neurological condition.

ELIGIBILITY:
Inclusion Criteria:

* Tracheostomy patient outside critical care
* Self-ventilating via a tracheostomy tube, independent of cuff status
* 18 years or older

Exclusion Criteria:

* Patients with tidal volume beyond recommended range (50-1000 ml)
* Dehydration
* Very heavy/excessive secretion from the lungs and airways (requiring more frequently tracheal suction, more than hourly suctioning)
* High oxygen need (FiO2 > 0.4)
* Acutely deteriorating patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of suctioning per day | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Times per day suctioning is required

SECONDARY OUTCOMES:
Time needed for suctioning | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Minutes per day of suctioning
Quality of secretion | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Amount and color of secretion
Quality of Life by EQ-5D-5L | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Patient reported, the descriptive system assesses health in five dimensions, from which a health state index score is calculated, range from 0 to 1, with higher scores indicating higher health utility
Use of TrachPhone | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  % of patients using TrachPhone/tolerating TrachPhone recorded by study specific questionnaire
Patient preference | Upon discharge from the hospital (on average after 3 weeks)
  % of patients (participants that were assigned to Arm 2) recorded by study specific questionnaire
Nurse and therapy team feedback | Upon discharge of the last participant, on average after 1 year
  Staff impression and preference measured by nurse survey
Nursing time regarding device use | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Minutes per day spent on device handling, recorded by nurse diary keeping, 3-day collection
Adherence to use of devices | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Hours of use of each humidification method, recorded by study specific questionnaire
Patient communication | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Communication by Therapy Outcome Measure for Voice Impairment (TOMS, score 0-5, higher score meaning no impairment)
Voice Quality | At Baseline, after 10 days, and every 10 days until discharge from hospital (on average after 3 weeks)
  Patient reported, for participants speaking, through study specific questionnaire
Patient mobility | Upon discharge of the last participant, on average after 1 year
  Staff perception of patient mobility and ease of transportation, measured though study specific questionnaires and nurse survey
Oxygen needs | At Baseline, T1 follow-up, and TX follow-ups every 10-14 days until discharge
  Weaning of oxygen time needed measured by peripheral oxygen saturation (%) recorded in patient charts. Only for monitoring reasons.
Adverse Events | Through study completion, an average of 1 year
  Any incidents reported throughout study duration

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Thomas, Dr, Principal Investigator — The Royal London Hospital, Barts Health NHS Trust
Locations (1):
- The Royal London Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No